CLINICAL TRIAL: NCT01208038
Title: Pilot Study: Evaluating the Effect of 300 Micrograms Testosterone Patches in Addition to Hormone Replacement Therapy on Arterial Compliance, Insulin Resistance and Sexual Desire.
Brief Title: Testosterone Patch's Effects on the Cardiovascular System and Libido
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Imperial College Healthcare NHS Trust (Other)
Collaborators: Royal Brompton & Harefield NHS Foundation Trust (Other); Chelsea and Westminster NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: CRO1646
Record Dates: First submitted 2010-09-22; First posted 2010-09-23 (Estimated); Results first posted 2020-01-02 (Actual); Last update posted 2020-01-02 (Actual); Status verified 2019-12

CONDITIONS: Hypoactive Sexual Desire Disorder
Keywords: Hypoactive sexual desire disorder
MeSH Terms: conditions — Sexual Dysfunctions, Psychological | interventions — Intrinsa

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Testosterone (Experimental): Testosterone transdermal patch 300micrograms, twice weekly for 12 weeks
  Interventions: Drug: Intrinsa Transdermal testosterone patch

INTERVENTIONS:
Drug: Intrinsa Transdermal testosterone patch — 300 microgram transdermal testosterone patch, applied twice weekly for 12 weeks
  Other Names: Intrinsa

SUMMARY:
The purpose of this study is to examine the effect of the testosterone patch, in addition to hormone replacement therapy (HRT), on blood vessel walls, insulin levels and sexual desire.

DETAILED DESCRIPTION:
A woman's ovaries produce the hormone testosterone during her reproductive life but testosterone levels decline with age or when the ovaries are removed. Testosterone has been associated with sexual desire in both men and women. Low testosterone is also believed to cause symptoms of low energy. Thus testosterone is increasingly used in hormone replacement regimens to restore libido and energy in postmenopausal women.

In the past testosterone has been administered orally or via subcutaneous implants. Recently testosterone patches have been licensed for treating low libido in postmenopausal women. The testosterone patches deliver a dose of testosterone equivalent to the levels produced by the ovary during a woman's early reproductive years.

Oral testosterone can lead to changes to insulin and cholesterol levels which increase the risk of heart disease. On the contrary, testosterone patches may reduce or avoid this risk. To date, trials have predominantly focused on safety data in terms of side effects and basic blood tests. Reviews of the safety of testosterone replacement have emphasised the need for improved safety data, especially in terms of cardiovascular risk.

The investigators hypothesis that transdermal testosterone, in addition to HRT, will have no adverse effects on blood vessel walls and insulin levels and that transdermal testosterone significantly improves sexuality and psychological well-being in postmenopausal women.

Trial design:

The investigators aim to recruit 20 postmenopausal women to wear the testosterone patch for 3 months in addition to their usual hormone replacement therapy.

There will be 3 study visits - a pre study visit, week 6 and week 12. At each visit the following procedures will be performed:

* Medical history and physical examination
* Blood sample - for hormone levels, lipids and insulin levels
* Blood vessel stiffness measurements This will be performed using a small ultrasound device at the wrist with blood pressure measured every 5 minutes.
* Endothelial function (function of your arterial wall) is measured using a blood pressure cuff on each arm and finger probes on one finger of each hand. The blood pressure cuff is inflated for 5 minutes and is then deflated quickly. The finger probes will record the readings throughout this study.
* Sexual satisfaction questionnaire

ELIGIBILITY:
Inclusion Criteria:

* healthy postmenopausal women
* 45 to 70 years of age
* on HRT and willing to continue the same HRT regimen for the next 6 months
* are in a stable relationship which was started at least 6 months ago
* continue on any concomitant medications without any change during the study
* give informed consent.

Exclusion Criteria:

* have dyspareunia
* have received testosterone implants within the last 12 months or other androgen therapy within the last 6 months
* have received any medications which may interfere with the study (SSRI, anti-androgens, PDE5 inhibitors, DHEA, SERMS)
* have a significant psychiatric disorder
* have a history of breast cancer
* have diabetes, thromboembolic disorders, cardiovascular disease, any condition affecting carbohydrate metabolism, uncontrolled hypertension and uncontrolled hyperlipidaemia
* are on tibolone (due to its androgenic effect).

Ages: 45 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2011-03 (Actual); Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nick Panay, MBBS, Principal Investigator — Imperial College Healthcare NHS Trust; John C Stevenson, MBBS, Principal Investigator — Royal Brompton and Harefield NHS Foundation Trust
Locations (3):
- United Kingdom (3):
  - Chelsea and Westminster Hospital, London
  - Queen Charlotte's and Chelsea Hospital, London
  - Royal Brompton Hospital, London

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Testosterone
Started | 22
Completed | 21 (Patient withdrew before commencing study drug)
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Population: Patient withdrew before baseline characteristics and starting study drug
Arm/Group | Testosterone
Number analyzed (Participants) | 21
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.0 (6.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21
  Male | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United Kingdom | 21
Augmentation Index [Mean (Standard Deviation); unit: percentage of Arterial stiffness] — Peripheral pressure waveforms were captured using radial artery application tonometry via the SphygmoCor apparatus (software version 8.0). The central pressure waveform was then derived from an averaged peripheral waveform using a validated, transfer function . The augmentation index (AIx), which gives a composite measure of wave reflection and systemic arterial stiffness can be calculated by analysis of the central waveform. Aix was defined as the difference between the first and second systolic peaks of the central pressure waveform, expressed as a percentage of the central pulse pressure.
  percentage of Arterial stiffness | 24.21 (10.70)
Reactive Hyperaemia Index [Mean (Standard Deviation); unit: Reactive hyperaemia index] — Reactive Hyperaemia Index (RHI) was calculated automatically by the EndoPAT 2000 computer algorithm from the ratio of pulse wave amplitude before and after ischaemia, compared to the control arm. Official reference values do not exists however a lower RHI (<2.0) is usually considered indicative of endothelial dysfunction.
  Reactive hyperaemia index | 1.79 (0.36)
Brief Profile of Female Sexual Function (B-PFSF) [Mean (Standard Deviation); unit: units on a scale] — Libido was assessed at each visit using the Brief profile of female sexual function (BPFSF), a validated self-administered questionnaire for identifying Hypoactive Sexual Desire Disorder (HSDD). The BPFSF is based on 7 questions. Each question is scored on a 6-point scale from 'always' to 'never'. A total score is calculated from a sum of all questions. Previous studies have identified a score of less than 20 as suggestive of HSDD.
  units on a scale | 15.3 (9.1)
Homeostatic Model Assessment of Insulin Resistance (HOMA-IR) [Mean (Standard Deviation); unit: units on a scale] — Blood samples were taken for fasting glucose and insulin levels. From these results, insulin resistance was then estimated using the updated homeostasis model assessment method for insulin resistance (HOMA-IR) computer algorithm. A higher HOMA-IR indicates a higher degree of insulin resistance. Typically a cutoff of HOMA-IR for identifying those with insulin resistance is 2.5.
  units on a scale | 0.78 (0.40)

OUTCOME MEASURES:

1. Primary Outcome: Arterial Compliance - Augmentation Index
Description: Peripheral pressure waveforms were captured using radial artery application tonometry via the SphygmoCor apparatus (AtCor Medical Ltd., Sydney, Australia; software version 8.0). The central (ascending aortic) pressure waveform was then derived from an averaged peripheral waveform using a validated, transfer function. The augmentation index (AIx), which gives a composite measure of wave reflection and systemic arterial stiffness can then be calculated by analysis of the central waveform. Aix was defined as the difference between the first and second systolic peaks of the central pressure waveform, expressed as a percentage of the central pulse pressure.
Time Frame: 12 weeks from baseline
Measure: Mean (95% Confidence Interval); unit: percentage of Arterial stiffness
Arm/Group | Testosterone
Number analyzed (Participants) | 21
percentage of Arterial stiffness | 1.067 [-3.85 to 1.72]

2. Primary Outcome: Endothelial Function
Description: Reactive Hyperaemia Index (RHI) was calculated automatically by the EndoPAT 2000 computer algorithm from the ratio of pulse wave amplitude before and after ischemia, compared to the control arm. Official reference values do not exist however a lower RHI (<2.0) is usually considered indicative of endothelial dysfunction.
Time Frame: 12 weeks from baseline
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Testosterone
Number analyzed (Participants) | 17
units on a scale | 0.06 [-0.19 to 0.31]

3. Secondary Outcome: Insulin Resistance - HOMA-IR
Description: Blood samples were taken for fasting glucose and insulin levels. From these results, insulin resistance was then estimated using the updated homeostasis model assessment method for insulin resistance (HOMA-IR) computer algorithm. A higher HOMA-IR indicates a higher degree of insulin resistance. Typically a cutoff of HOMA-IR for identifying those with insulin resistance is 2.5.
Time Frame: 12 weeks from baseline
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Testosterone
Number analyzed (Participants) | 21
units on a scale | 0.106 [-0.20 to 0.41]

4. Secondary Outcome: Libido - B-PFSF Score
Description: Libido was assessed at each visit using the Brief profile of female sexual function (BPFSF), a validated self-administered questionnaire for identifying Hypoactive Sexual Desire Disorder (HSDD). The BPFSF is based on 7 questions. Each question is scored on a 6-point scale from 'always' to 'never'. A total score is total score ranging from 0 to 35. Previous studies have identified a score of less than 20 as suggestive of HSDD.
Time Frame: 12 weeks from baseline
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Testosterone
Number analyzed (Participants) | 21
units on a scale | 5.05 [2.63 to 7.46]

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | Testosterone
All-Cause Mortality (participants affected / at risk) | 0/21
Serious Adverse Events (participants affected / at risk) | 0/21
Other Adverse Events (participants affected / at risk) | 7/21
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Testosterone (N=21)
Skin irritation (Skin and subcutaneous tissue disorders) | 4
Increased facial hair (Endocrine disorders) | 2
Acne (Skin and subcutaneous tissue disorders) | 1
per vagina spotting (Reproductive system and breast disorders) | 1
Blepharitis (Eye disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No